CLINICAL TRIAL: NCT07217925
Title: Exploring the Influence of Neurofeedback on the Well-Being of People With Symptoms of Obsessive Compulsive Disorder and Post-traumatic Stress Symptoms
Brief Title: Neurofeedback and Well-Being Among People With Co-Occurring Obsessive Compulsive Disorder and Post-traumatic Stress Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Lisa S. Panisch, PhD, MSW, Assistant Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-25-07-7918
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Well-Being, Psychological; Mood Disturbance; Emotional Regulation; Dissociation; Post Traumatic Stress Symptoms
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation; Dissociative Disorders | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neurofeedback Training (Other): Participants in the Neurofeedback Training group will complete per-training, post-training, and post-training follow-up self-report surveys assessing overall well-being, symptoms of obsessive compulsive disorder, post-traumatic stress, OCD, dissociation and other trauma-related mental health symptoms, emotional regulation, etc. Participants in this group will all be on a wait list to receive obsessive compulsive disorder-specific psychotherapy at a local outpatient therapy clinic that specializes in the treatment of anxiety and obsessive compulsive disorders. All participants will demonstrate clinically significant post-traumatic stress symptoms and have a self-reported diagnosis of obsessive compulsive disorder.
  Interventions: Device: Neuroptimal (Zengar, Inc.) Neurofeedback

INTERVENTIONS:
Device: Neuroptimal (Zengar, Inc.) Neurofeedback — Participants in the Neurofeedback Training group will complete a total of 8 training sessions (1-2 sessions a week, each session lasting approximately 34 minutes) within a 3 month time span, using the Neuroptimal (Zengar, Inc.) neurofeedback device.

SUMMARY:
The proposed study will collect novel data evaluating the feasibility of a neurofeedback training program delivered to prospective clients with a history of clinically concerning trauma-related mental health symptoms who are on a wait list to receive obsessive compulsive disorder-specific psychotherapy at an outpatient mental health clinic. This study will evaluate the influence of neurofeedback training on participant's overall sense of well-being, and additionally, whether any enhanced well-being is subsequently associated with positive changes in symptoms of obsessive compulsive disorder, post-traumatic stress, dissociation and other trauma-related mental health symptoms, emotional regulation, etc.

ELIGIBILITY:
Inclusion Criteria:

1. being a client placed on the clinic waitlist to receive exposure-response prevention for OCD symptoms at the Anxiety and OCD Treatment Center of Ann Arbor, in Ann Arbor, MI.
2. having self-reported symptoms of OCD;
3. having post-traumatic stress symptoms as indicated by a score of 3 or higher on the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) screening measure;
4. being age 18+.
5. being a citizen of the United States of America -

Exclusion Criteria:

1. a lifetime history of significant untreated mental illness (not currently treated schizophrenia, schizoaffective disorder, bipolar disorder, or substance use disorder) or neurological or pervasive developmental disorder;
2. a documented history of epilepsy;
3. lifetime history of any head injury with loss of consciousness;
4. current exposure domestic or intimate partner violence or otherwise state that their current living conditions are unsafe;
5. current experiences of psychosis or suicidality within the last six months;
6. currently taking, or in the past month has taken benzodiazepines, narcotic drugs, or cannabis;
7. currently pregnant
8. engagement in self-harming behaviors in the last 3 months that required medical attention;
9. lack of competence to understand or consent to the study procedures;
10. lack of fluency in written and spoken English. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders, Fith Edition (PTSD Checklist for DSM-5 - Standard). | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  This measure evaluates symptoms of post-traumatic stress. Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.
Dissociative Symptoms Scale (DSS) | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  This 20-item measure evaluates moderate to severe levels of dissociative symptoms in four main domains: depersonalization, derealization, gaps in awareness or memory, and dissociative reexperiencing symptoms. Scores range from 0-80, with higher scores indicating worse outcomes.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS; with Checklist) | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  10-item measure evaluating severity of obsessive compulsive symptoms, with an accompanying checklist of symptom types. Scores range from 0-40 with higher scores indicating worse outcomes. Symptoms on the checklist are categorized, and indicate different OCD symptom clusters or sub-types that respondents may experience.
Difficulties in Emotion Regulation Scale (DERS) | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  36-item measure evaluating challenges with emotional regulation. Scores range from 36-180, with higher scores indicating worse outcomes.
The World Health Organization-Five Well-Being Index (WHO-5) | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  5-item measure evaluating overall well-being. Scores range from 0-25, with higher scores indicating better outcomes.
Patient Health Questionnaire - 8 (PHQ-8) | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  8-item measure evaluating depressive symptoms. Scores range from 0-24, with higher scores indicating worse outcomes.
GAD-7 | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  7-item measure evaluating anxiety symptoms. Scores range from 0-21, with higher scores indicating worse outcomes.
Everyday Discrimination Scale | The measure will be administered three intervals: 1) per-training, at the beginning of the study, 2) post-training, between 2-3 months later, following the completion of the training phase, 3) as a follow-up, 3 months after the post-training interval.
  9-item measure evaluating experiences of discrimination. Scores range from 9-54, with higher scores indicating more frequent experiences of discrimination.